CLINICAL TRIAL: NCT01544764
Title: Examining Adolescent Assessment, Feedback, Incentive, and Exchange (AFIX)
Brief Title: Examining Adolescent Assessment, Feedback, Incentive, and Exchange (AFIX) in North Carolina
Acronym: AFIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Division of Public Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011-3
Record Dates: First submitted 2012-02-24; First posted 2012-03-06 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Adolescent Health Services; Immunization
Keywords: Diphtheria-Tetanus-Pertussis Vaccine; Measles-Mumps-Rubella Vaccine; Meningococcal Vaccines; Hepatitis B Vaccines; Chickenpox Vaccine; Papillomavirus Vaccines
MeSH Terms: conditions — Hepatitis B | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): This arm includes 30 health centers in North Carolina with at least 200 adolescent (age 11-18) patients. Practices in this arm were randomly assigned to receive no AFIX visit.
- AFIX In-Person Visit (Experimental): This arm includes 30 health centers in North Carolina with at least 200 adolescent (age 11-18) patients. These practices received an in-person AFIX visit from a North Carolina Immunization Branch employee.
  Intervention:
  Other: Assessment , Feedback, Incentives, and eXchange Program
  Interventions: Other: Assessment , Feedback, Incentives, and eXchange Program
- AFIX Webinar Visit (Experimental): This arm includes 31 health centers in North Carolina with at least 200 adolescent (age 11-18) patients. These practices received a webinar during which a North Carolina Immunization Branch employee completed the components of an AFIX visit.
  Intervention:
  Other: Assessment , Feedback, Incentives, and eXchange Program
  Interventions: Other: Assessment , Feedback, Incentives, and eXchange Program

INTERVENTIONS:
Other: Assessment , Feedback, Incentives, and eXchange Program — The NC Immunization Branch uses Adolescent AFIX (Assessment, Feedback, Incentives and eXchange) Program, a quality improvement strategy developed by the CDC to improve the immunization practices and vaccination coverage levels of public and private health care providers. It has four main components: 1) Assessment of a provider's current immunization practices and vaccination levels, 2) Feedback of the assessment results and strategies to improve coverage levels, 3) Incentives to improve coverage levels, and 4) eXchange of information and resources necessary to facilitate improvement.
  Arms: AFIX In-Person Visit; AFIX Webinar Visit

SUMMARY:
The North Carolina Immunization Branch will evaluate the use of the CDC program to improve adolescent vaccination practices (called Assessment, Feedback, Incentives, and eXchanges, or AFIX). This evaluation is the first of its kind in the nation and may have a profound impact on prevention.

AFIX has four major components: 1) Assessment of a provider's current immunization practices and vaccination levels, 2) Feedback of the assessment results and strategies to improve coverage levels, 3) Incentives to improve coverage levels, and 4) eXchange of information and resources necessary to facilitate improvement.

This program will evaluate the effectiveness of AFIX visits on affecting provider practices to increase adolescent (age 11-18) immunization. Visits include discussion of that practice's immunization rates and strategies for improving rates. The investigators will compare the changes, from baseline to 5 months, in immunization for practices receiving virtual visits (webinars), in-person visits, and no visits (control group). Thirty practices will be randomly assigned to each intervention type. The main outcomes of this study are practice-wide uptake rates of several adolescent vaccines (Tdap, HPV, and MCV4) as well as pre- and post-AFIX visit surveys focusing on recall tactics utilized by each practice. Data will be collected on practices with at least 200 adolescent patients (note: there is no patient-level data collected in this study).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric and/or family practices participating in the North Carolina Immunization Program
* A minimum of 200 active adolescent patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in Vaccination Rate: HPV vaccine initiation among 11-12 year olds | Baseline and 5 months follow-up
  We will gather practice-specific rates of coverage for adolescents (age 11-12) for the first dose of human papillomavirus (HPV) vaccine at baseline and 5 months follow-up.

SECONDARY OUTCOMES:
Change in Vaccination Rate: HPV vaccine initiation among 13-18 year olds | Baseline and 5 months follow-up
  We will gather practice-specific rates of coverage for adolescents (age 13-18) for the first dose of human papillomavirus (HPV) vaccine at baseline and 5 months follow-up.
Change in Vaccination Rate: Tdap vaccine among 11-12 year olds | Baseline and 5 months follow-up
  We will gather practice-specific rates of coverage for adolescents (age 11-12) for tetanus, diphtheria, and pertussis booster (Tdap) at baseline and 5 months follow-up.
Change in Vaccination Rate: Tdap vaccine among 13-18 year olds | Baseline and 5 months follow-up
  We will gather practice-specific rates of coverage for adolescents (age 13-18) for tetanus, diphtheria, and pertussis booster (Tdap) at baseline and 5 months follow-up.
Change in Vaccination Rate: Meningitis vaccine among 11-12 year olds | Baseline and 5 months follow-up
  We will gather practice-specific rates of coverage for adolescents (age 11-12) for meningococcal conjugate (i.e., meningitis vaccine) at baseline and 5 months follow-up.
Change in Vaccination Rate: Meningitis vaccine among 13-18 year olds | Baseline and 5 months follow-up
  We will gather practice-specific rates of coverage for adolescents (age 13-18) for meningococcal conjugate (i.e., meningitis vaccine) at baseline and 5 months follow-up.
Change in Vaccination Rate: HPV vaccine completion among 11-12 year olds | Baseline and 5 months follow-up
  We will gather practice-specific rates of coverage for adolescents (age 11-12) for the third and final dose of human papillomavirus (HPV) vaccine at baseline and 5 months follow-up.
Change in Vaccination Rate: HPV vaccine completion among 13-18 year olds | Baseline and 5 months follow-up
  We will gather practice-specific rates of coverage for adolescents (age 13-18) for the third and final dose of human papillomavirus (HPV) vaccine at baseline and 5 months follow-up.

OTHER OUTCOMES:
Change in Vaccination Rate: MMR among 11-12 year olds | Baseline and 5 months follow-up
  We will gather practice-specific rates of coverage for adolescents (ages 11-12) for measles, mumps, and rubella (MMR) vaccine at baseline and 5 months follow-up. This is a childhood vaccine that is not targeted for adolescents; however the intervention may impact MMR coverage.
Change in Vaccination Rate: MMR among 13-18 year olds | Baseline and 5 months follow-up
  We will gather practice-specific rates of coverage for adolescents (ages 13-18) for measles, mumps, and rubella (MMR) vaccine at baseline and 5 months follow-up. This is a childhood vaccine that is not targeted for adolescents; however the intervention may impact MMR coverage.
Change in Vaccination Rate: Hepatitis B vaccine among 11-12 year olds | Baseline and 5 months follow-up
  We will gather practice-specific rates of coverage for adolescents (ages 11-12) for hepatitis B vaccine at baseline and 5 months follow-up. This is a childhood vaccine that is not targeted for adolescents; however the intervention may impact hepatitis B vaccine coverage.
Change in Vaccination Rate: Hepatitis B vaccine among 13-18 year olds | Baseline and 5 months follow-up
  We will gather practice-specific rates of coverage for adolescents (ages 13-18) for hepatitis B vaccine at baseline and 5 months follow-up. This is a childhood vaccine that is not targeted for adolescents; however the intervention may impact hepatitis B vaccine coverage.
Change in Vaccination Rate: Varicella vaccine among 11-12 year olds | Baseline and 5 months follow-up
  We will gather practice-specific rates of coverage for adolescents (ages 11-12) for varicella vaccine at baseline and 5 months follow-up. This is a childhood vaccine that is not targeted for adolescents; however the intervention may impact varicella vaccine coverage.
Change in Vaccination Rate: Varicella vaccine among 13-18 year olds | Baseline and 5 months follow-up
  We will gather practice-specific rates of coverage for adolescents (ages 13-18) for varicella vaccine at baseline and 5 months follow-up. This is a childhood vaccine that is not targeted for adolescents; however the intervention may impact varicella vaccine coverage.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Dayton, MA, Principal Investigator — DPH/WCH/Immunization; Amy Grimshaw, MS, MSW, Principal Investigator — DPH/WCH/Immunization; Noel T Brewer, PhD, Study Director — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Cervical Cancer-Free North Carolina, Chapel Hill, North Carolina
  - North Carolina Immunization Branch, Raleigh, North Carolina

REFERENCES:
- [Derived] Gilkey MB, Dayton AM, Moss JL, Sparks AC, Grimshaw AH, Bowling JM, Brewer NT. Increasing provision of adolescent vaccines in primary care: a randomized controlled trial. Pediatrics. 2014 Aug;134(2):e346-53. doi: 10.1542/peds.2013-4257. Epub 2014 Jul 7. PMID 25002671
- [Derived] Gilkey MB, Moss JL, Roberts AJ, Dayton AM, Grimshaw AH, Brewer NT. Comparing in-person and webinar delivery of an immunization quality improvement program: a process evaluation of the adolescent AFIX trial. Implement Sci. 2014 Feb 18;9:21. doi: 10.1186/1748-5908-9-21. PMID 24533515